CLINICAL TRIAL: NCT06698432
Title: Prognostic Implications of Stress Hyperglycemia Ratio for the Prognosis of Coronary Microvascular Dysfunction in Patients with Chronic Coronary Syndrome
Brief Title: SHR Predicts CMD in Patients with CCS
Acronym: SHR-CMD-CCS
Status: Completed | Type: Observational
Sponsor: Ya-Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: SHR-CMD-CCS
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Coronary Microvascular Dysfunction (CMD); Index of Microvascular Resistance; Chronic Coronary Syndrome; Prognosis
Keywords: Coronary Microvascular Dysfunction (CMD); Coronary angiography-derived index of microvascular resistance; Chronic coronary syndrome; Stress hyperglycemia ratio; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CMD: Microvascular function was assessed using caIMR, CMD was identified with caIMR>25U, in line with prior research.
  Interventions: Device: caIMR
- non-CMD: Microvascular function was assessed using caIMR, non-CMD was identified with caIMR≤25U, in line with prior research.
  Interventions: Device: caIMR

INTERVENTIONS:
Device: caIMR — Coronary angiography-derived IMR (caIMR) is a novel and accurate alternative that can enable the assessment of coronary microvascular function easier, and more efficiently and does not require pressure wire or adenosine.

SUMMARY:
SHR exerts a significant influence in numerous cardiovascular diseases, including MINOCA (myocardial infarction with non - obstructive coronary arteries), HFpEF (heart failure with preserved ejection fraction), and CAD (coronary artery disease). It thereby demonstrates its predictive capacity regarding survival risk and its value in risk-stratification procedures. To date, no studies have specifically investigated the prognostic implications of the stress hyperglycemia ratio (SHR) in CMD patients with CCS, highlighting the need for further research. Therefore, this study seeks to evaluate the predictive value of the stress hyperglycemia ratio (SHR) in CMD patients with CCS, and to elucidate its clinical relevance and significance, which remain poorly understood in this patient cohort.

DETAILED DESCRIPTION:
Coronary artery disease (CAD), a cardiovascular disorder precipitated by the atherosclerotic narrowing or occlusion of the coronary arteries, culminates in myocardial ischemia, hypoxia, or necrosis. As one of the foremost causes of morbidity and mortality worldwide, CAD represents an escalating public health concern. Chronic coronary syndrome (CCS) refers to the stable, long-term clinical manifestations of coronary artery disease (CAD), representing a progressive and sustained phase of the condition. Coronary microvascular dysfunction (CMD) is characterized by alterations in the structure and function of the coronary microcirculation, a condition frequently encountered in clinical practice. The presence of CMD, particularly when associated with atherosclerosis, may exacerbate myocardial ischemia in patients with chronic coronary syndrome (CCS). CMD is prevalent across a broad range of cardiovascular conditions, including heart failure with preserved ejection fraction (HFpEF), Takotsubo syndrome (TTS), acute coronary syndrome (ACS), myocardial infarction with non-obstructive coronary arteries (MINOCA), and CCS. It plays a pivotal role in the pathophysiology and prognosis of these diseases. Substantial evidence indicates that coronary microvascular dysfunction (CMD) is prevalent in patients with chronic coronary syndrome (CCS) and is closely linked to the pathogenesis and unfavorable prognosis of the condition. Therefore, the diagnosis of CMD carries significant implications for the management of CCS patients and the prevention of adverse outcomes.

The molecular mechanisms of CMD are not yet fully understood, but impaired pathologic dilation or increased constriction of coronary microvessels due to oxidative stress and inflammatory responses are thought to be the vital causative mechanisms of CMD.Studies have demonstrated that hyperglycemic states play a crucial role in CMD by altering the oxygen demand of cardiomyocytes, which leads to abnormal vascular regulation.Stress-induced hyperglycemia may aggravate coronary microvascular dysfunction (CMD) through mechanisms such as the induction of endothelial dysfunction and the promotion of oxidative stress, thereby contributing to adverse outcomes. Acute hyperglycemia, often undetected due to the lack of precise and effective monitoring methods, may arise from either pre-existing chronic hyperglycemia or acute physiological stress, leading to a transient increase in blood glucose levels upon hospital admission. In these instances, the stress hyperglycemia ratio (SHR) has been proposed as a novel marker to more accurately reflect the acute hyperglycemic state. The SHR is defined as the ratio of the blood glucose level at admission to the estimated average chronic glycemic value. SHR exerts a significant influence in numerous cardiovascular diseases, including MINOCA (myocardial infarction with non - obstructive coronary arteries), HFpEF (heart failure with preserved ejection fraction), and CAD (coronary artery disease). It thereby demonstrates its predictive capacity regarding survival risk and its value in risk-stratification procedures. To date, no studies have specifically investigated the prognostic implications of the stress hyperglycemia ratio (SHR) in CMD patients with CCS, highlighting the need for further research. Therefore, this study seeks to evaluate the predictive value of the stress hyperglycemia ratio (SHR) in CMD patients with CCS, and to elucidate its clinical relevance and significance, which remain poorly understood in this patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* (1)Patients aged over 18 years (2)Patients diagnosed as suspected or established CCS[PMID: 39210710]who subsequently underwent coronary angiography (CAG).

Exclusion Criteria:

- (1)A left ventricular ejection fraction (LVEF) lower than 35% (2)Recent occurrence of myocardial infarction (MI) (3)Severe hepatic or renal dysfunction (4)The existence of malignancy (5)Post-coronary artery bypass graft surgery (CABG) (6)Being in a current state of pregnancy (7)Incomplete data of SHR, (8)Non-adherence to follow-up protocols (9)Other life-threatening diseases that significantly impact long-term survival.

(10) Suboptimal quality of angiography images, evident vascular overlap, distortion of the investigated artery or low contrast opacification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This single-center retrospective observational study were implemented in Shanghai Tenth People's Hospital spanning from June 2015 to June 2019. Our investigation received the endorsement of the Ethical Review Board of Shanghai Tenth People's Hospital and was carried out in line with the Helsinki Declaration. Each patient involved in this study was required to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac events (MACE) | Follow-up was conducted over a mean 43-month period through telephone calls, hospital records, and outpatient visits by trained physicians at Shanghai Tenth People's Hospital
  We defined major adverse cardiac events (MACE) as the primary clinical endpoint of present investigation, which was a combination of following conditions: (1) Cardiac death: demise caused by malignant arrhythmia, acute MI, heart failure, or other cardiac diseases; (2) Ischemia-driven revascularization: revascularization due to recurrent angina or a positive cardiac ischemia test; (3) Nonfatal MI: presence of positive cardiac biomarkers along with typical myocardial ischemia symptoms or electrocardiogram dynamic changes; (4) Heart failure: clinical symptoms such as dyspnea, fatigue, etc., accompanied by positive evidence from echocardiography, BNP/NT-proBNP measurement, and cardiac function assessment; (5) Nonfatal stroke: acute cerebral infarction diagnosed by typical clinical symptoms or imaging examination.

IPD SHARING:
Plan to Share IPD: No